CLINICAL TRIAL: NCT03527316
Title: Effect of MDMA (Serotonin Release) on Fear Extinction
Brief Title: Effect of Methylenedioxymethamphetamine (MDMA) (Serotonin Release) on Fear Extinction
Acronym: MFE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BASEC 2017-01947
Record Dates: First submitted 2018-05-04; First posted 2018-05-17 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Healthy
MeSH Terms: interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MDMA, Placebo (Experimental): Cross-over within-subjects design with both treatment conditions, separated by a wash-out phase
  Interventions: Drug: MDMA; Drug: Placebo
- Placebo, MDMA (Experimental): Cross-over within-subjects design with both treatment conditions, separated by a wash-out phase
  Interventions: Drug: MDMA; Drug: Placebo

INTERVENTIONS:
Drug: MDMA — 125 mg MDMA per os, single dose
  Other Names: 3,4-Methylenedioxymethamphetamine
Drug: Placebo — Capsules containing mannitol looking identical to the other drugs.

SUMMARY:
Serotonin and oxytocin play a role in fear conditioning and fear extinction learning, psychological processes that are critically involved in psychiatric disorders such as posttraumatic stress disorder (PTSD). Specifically, administration of oxytocin has been shown to facilitate fear extinction in humans. Similarly, substances that release serotonin and oxytocin such as MDMA have been shown to enhance the extinction of fear memory in animals. However, there are no data on the effects of MDMA on fear extinction in humans. Therefore, the primary aim of this study is to investigate the role of acute serotonin release in the effects of fear extinction. MDMA will be used as pharmacological tool to induce serotonin release in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 18 and 50 years.
* Understanding of the German language.
* Understanding the procedures and the risks associated with the study.
* Participants must be willing to adhere to the protocol and sign the consent form.
* Participants must be willing to refrain from taking illicit psychoactive substances during the study.
* Participants must be willing to drink only alcohol-free liquids and no coffee, black or green tea, or energy drink after midnight of the evening before the study session, as well as during the study day.
* Participants must be willing not to drive a traffic vehicle or to operate machines within 48 h after substance administration.
* Body mass index 18-29 kg/m2.

Exclusion Criteria:

* Chronic or acute medical condition
* Hypertension (>140/90 mmHg) or hypotension (SBP<85 mmHg)
* Current or previous major psychiatric disorder
* Psychotic disorder in first-degree relatives
* Illicit substance use (with the exception of cannabis) of more than 5 times or any time within the previous month.
* Participation in another clinical trial (currently or within the last 30 days)
* Use of medications that may interfere with the effects of the study medications (any psychiatric medications)
* Tobacco smoking (>10 cigarettes/day)
* Consumption of alcoholic standard drinks (>10/week or >120 g ethanol/week)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Fear extinction measured by Skin conductance response | 12 months
  a) Skin conductance response to conditioned stimuli
Fear extinction measured by Fear-potentiated startle | 12 months
  b) Fear-potentiated startle to conditioned stimuli

SECONDARY OUTCOMES:
Plasma concentration of Oxytocin | 12 months
Subjective effects measured by Visual analog scales | 12 months
  Visual analog scales, 0-100, 0 for 'not at all' and 100 for 'extremely'
Autonomic effects measured by Blood pressure | 12 months
  Autonomic effects measured by vital signs
Autonomic effects measured by Hearth rate | 12 months
  Autonomic effects measured by vital signs
Autonomic effects measured by Body temperature | 12 months
  Autonomic effects measured by vital signs
Subjective effects measured by State-trait anxiety inventory for state (STAI-S) | 12 months
Plasma concentration of MDMA | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, MAS, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Clinical Pharmacology & Toxicology, University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vizeli P, Straumann I, Duthaler U, Varghese N, Eckert A, Paulus MP, Risbrough V, Liechti ME. Effects of 3,4-Methylenedioxymethamphetamine on Conditioned Fear Extinction and Retention in a Crossover Study in Healthy Subjects. Front Pharmacol. 2022 Jul 13;13:906639. doi: 10.3389/fphar.2022.906639. eCollection 2022. PMID 35910354